CLINICAL TRIAL: NCT04251546
Title: Prediction Model fo Screening and Diagnosis of Prostate Cancer in PSA Gray Zone Based on Serum PHI Combined With TPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-20-002
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; PSA
Keywords: Prostate Cancer; PSA; PHI; ultrasound; TPV
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients with suspected prostate cancer with a PSA test value of 4-10 ng / mL
  Interventions: Diagnostic Test: p2PSA; Diagnostic Test: Ultrasonic parameters; Diagnostic Test: Transperineal prostate biopsy

INTERVENTIONS:
Diagnostic Test: p2PSA — p2PSA test(for calculation of PHI)
Diagnostic Test: Ultrasonic parameters — Ultrasonic parameters(TPV)
Diagnostic Test: Transperineal prostate biopsy — Transperineal prostate biopsy for confirmation of prostate cancer or benign disease

SUMMARY:
Prostate cancer (PCa) is a high incidence tumor of elderly men. In recent years, its incidence has rapidly increased in China. Serological examination of prostate-specific antigen (PSA) is particularly important in the early diagnosis of PCa, but its specificity is lower in gray areas with PSA between 4-10 ng / ml. Proposition of prostate health index (PHI) strengthens the specificity of PSA gray area prostate cancer diagnosis, but the composition of the index only relies on serological examination, neglects imaging indicators, and cannot be comprehensively evaluated. Based on the preliminary basis of PHI research in the undergraduate department, combined with ultrasound imaging indicators of total prostate volume (TPV), this research group prospectively analyzed the efficacy of PHI combined with TPV to predict prostate cancer in patients with PSA gray areas, and established an improved version of PHI-TPV combination. The prediction model mPHI assesses the sensitivity of the new model to predict the risk of prostate cancer in the Chinese population, provides data support for puncture decisions of middle-aged and elderly male patients in the gray area of PSA in China, and provides reference and guidance for the individualized prevention and treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient> 45 years of age
2. Abnormal serum PSA
3. Prostate nodules found by DRE
4. Abnormal MRI or TRUS finding

Exclusion Criteria:

1. Incomplete medical history
2. Poor quality of serum samples
3. Bacterial acute prostatitis diagnosed within 3 months before biopsy 4.5α reductase inhibitors, anabolic steroids, or antiandrogen drugs taken within 12 months before biopsy

5.Previous prostate biopsy history.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study selected patients with suspected prostate cancer in the Department of Urology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine from May 2019 to May 2022, and had a PSA test value of 4-10 ng / mL.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-04 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological confirmed diagnosis of prostate cancer or benign prostatic diseases | 2019/05/01-2021/05/30
  Pathological confirmed diagnosis by transrectal ultrasound guided prostate biopsy (12 needles) according to a standardized protocol. If a suspicious low-density nodule is found during the ultrasound, biopsy to the nodule can be added. Place the prostate biopsy specimen in a 10% Formalin's specimen bag. The specimens were processed and evaluated by the Pathology Department of Xinhua Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen H, Qian Y, Wu Y, Shi B, Zhou J, Qu F, Gu Z, Ding J, Yu Y. Modified Prostate Health Index Density Significantly Improves Clinically Significant Prostate Cancer (csPCa) Detection. Front Oncol. 2022 Apr 7;12:864111. doi: 10.3389/fonc.2022.864111. eCollection 2022. PMID 35463344